CLINICAL TRIAL: NCT04460378
Title: Exposure Initializes Therapy - Treatment Of Homebound Patients Extended
Acronym: ExITTOHoPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Humboldt-Universität zu Berlin (Other); Stiftung Deutsche Klassenlotterie Berlin (Unknown)
Responsible Party: Principal Investigator, Dr. Jens Plag, Dr. med. Jens Plag, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChariteAmb
Record Dates: First submitted 2018-03-22; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Agoraphobia
MeSH Terms: conditions — Agoraphobia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: repeated measure of a single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Therapy (Experimental): Manualized Cognitive Behavioral Therapy starting at the patients' home.
  Interventions: Behavioral: cognitive behavioral therapy

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — cognitive behavioral therapy with Focus on guided exposure

SUMMARY:
Cognitive behavioral treatment of homebound patients with severe agoraphobia.

DETAILED DESCRIPTION:
Homebound patients with severe agoraphobia are treated with an exposure focussed cognitive behavioral therapy. The treatment begins at home. With a quick onset of guided exposure, patients get the possibility to develope the capability to reach the regular Treatment Location on their own very rapidly.

ELIGIBILITY:
Inclusion Criteria:

* agoraphobia with/without Panic disorder

Exclusion Criteria:

* psychotic disorders
* bipolar disorders
* acute substance dependency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
MI | Change from baseline to 4th psychotherapy session (+42 days) and change from baseline to the 9th psychotherapy session (+60 days) and change from baseline to follow up (+98 days)
  Mobility Inventory

SECONDARY OUTCOMES:
AKF | Change from baseline to 4th psychotherapy session (+42 days) and change from baseline to the 9th psychotherapy session (+60 days) and change from baseline to follow up (+98 days)
  Angst-Kontroll-Fragebogen (anxiety control)
ASI | Change from baseline to 4th psychotherapy session (+42 days) and change from baseline to the 9th psychotherapy session (+60 days) and change from baseline to follow up (+98 days)
  Angstsensitivität (anxiety sensitivity)
NEO-FFI | Change from baseline to 4th psychotherapy session (+42 days) and change from baseline to the 9th psychotherapy session (+60 days) and change from baseline to follow up (+98 days)
  Persönlichkeitsfragebogen (personality inventory)
PSQ 20 | Change from baseline to 4th psychotherapy session (+42 days) and change from baseline to the 9th psychotherapy session (+60 days) and change from baseline to follow up (+98 days)
  perceived stress questionnaire
rs 13 | Change from baseline to 4th psychotherapy session (+42 days) and change from baseline to the 9th psychotherapy session (+60 days) and change from baseline to follow up (+98 days)
  Resilienzskala (resilience scale)
SWE | Change from baseline to 4th psychotherapy session (+42 days) and change from baseline to the 9th psychotherapy session (+60 days) and change from baseline to follow up (+98 days)
  Selbstwirksamkeitsfragebogen (self-efficacy questionnaire)
UI18 | Change from baseline to 4th psychotherapy session (+42 days) and change from baseline to the 9th psychotherapy session (+60 days) and change from baseline to follow up (+98 days)
  Unsicherheitsintoleranz Fragebogen (intolerance of uncertainty questionnaire)
EQ-5D | Change from baseline to 4th psychotherapy session (+42 days) and change from baseline to the 9th psychotherapy session (+60 days) and change from baseline to follow up (+98 days)
  life quality questionnaire
AAQ II | Change from baseline to 4th psychotherapy session (+42 days) and change from baseline to the 9th psychotherapy session (+60 days) and change from baseline to follow up (+98 days)
  Acceptance and Action questionnaire
ACQ | Change from baseline to 4th psychotherapy session (+42 days) and change from baseline to the 9th psychotherapy session (+60 days) and change from baseline to follow up (+98 days)
  Agoraphobic cognition questionnaire
BSQ | Change from baseline to 4th psychotherapy session (+42 days) and change from baseline to the 9th psychotherapy session (+60 days) and change from baseline to follow up (+98 days)
  Bosy Sensation Questionnaire
BDI II | Change from baseline to 4th psychotherapy session (+42 days) and change from baseline to the 9th psychotherapy session (+60 days) and change from baseline to follow up (+98 days)
  Beck Depression inventory II
alpha-amylase | change from baseline to follow up (+98 days)
  daily profile of salivary alpha amylase
cortisol | change from baseline to follow up (+98 days)
  daily profile of salivary cortisol
PAS | Change from baseline to 4th psychotherapy session (+42 days) and change from baseline to the 9th psychotherapy session (+60 days) and change from baseline to follow up (+98 days)
  Panik- und Agoraphobie-Skala (Panic and agoraphobia scale)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Plag, MD, Study Chair — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided